CLINICAL TRIAL: NCT01550471
Title: A Study Evaluating the Effect of Omnaris Nasal Spray 200 mcg QD & Alvesco Inhalation Aerosol 80 BID vs Beconase AQ Nasal Spray 168 mcg BID & QVAR Inhalation Aerosol 40 mcg BID vs Placebo Nasal Spray QD & Placebo Inhalation Aerosol BID on Short Term Growth in Pediatric Subjects With Mild Asthma & Allergic Rhinitis
Brief Title: Sunovion Growth Study Pediatric Subjects With Mild Asthma & Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Deborah Gentile, Principal Investigator, West Penn Allegheny Health System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RC#5401
Record Dates: First submitted 2012-02-19; First posted 2012-03-12 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: Mild asthma and allergic rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — ciclesonide; Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 Treatment Sequence-A and O, Q and B, P and P (Experimental): Period 2-Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD Period 4-QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID Period 6-Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID
  Interventions: Drug: Alvesco/Omnaris, QVAR/Beconase, Placebo/Placebo
- 2 Treatment Sequence-A and O, P and P, Q and B (Experimental): Period 2-Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD Period 4-Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID Period 6-QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID
  Interventions: Drug: Alvesco/Omnaris, Placebo/Placebo, QVAR/Beconase
- 3 Treatment Sequence-Q and B, A and O, P and P (Experimental): Period 2-QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID Period 4-Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD Period 6-Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID
  Interventions: Drug: QVAR/Beconase, Alvesco/Omnaris, Placebo/Placebo
- 4 Treatment Sequence-Q and B, P and P, A and O (Experimental): Period 2-QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID Period 4-Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID Period 6-Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD
  Interventions: Drug: QVAR/Beconase, Placebo/Placebo, Alvesco/Omnaris
- 5 Treatment Sequence-P and P, A and O, Q and B (Experimental): Period 2-Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID Period 4-Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD Period 6-QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID
  Interventions: Drug: Placebo/Placebo, Alvesco/Omnaris, QVAR/Beconase
- 6 Treatment Sequence-P and P, Q and B, A and O (Experimental): Period 2-Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID Period 4-QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID Period 6-Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD
  Interventions: Drug: Placebo/Placebo, QVAR/Beconase, Alvesco/Omnaris

INTERVENTIONS:
Drug: Alvesco/Omnaris, QVAR/Beconase, Placebo/Placebo — Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID Placebo Nasal Spray QD/Placebo Inhalation Aerosol BID
  Other Names: Ciclesonide, Beclomethasone, Placebo
  Arms: 1 Treatment Sequence-A and O, Q and B, P and P
Drug: Alvesco/Omnaris, Placebo/Placebo, QVAR/Beconase — Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD, Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID, QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID
  Other Names: Ciclesonide, Placebo, Beclomethasone
  Arms: 2 Treatment Sequence-A and O, P and P, Q and B
Drug: QVAR/Beconase, Alvesco/Omnaris, Placebo/Placebo — QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID, Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD, Placebo Nasal Spray QD/Placebo Inhalation Aerosol BID
  Other Names: Beclomethasone, Ciclesonide, Placebo
  Arms: 3 Treatment Sequence-Q and B, A and O, P and P
Drug: QVAR/Beconase, Placebo/Placebo, Alvesco/Omnaris — QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID, Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID, Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD
  Other Names: Beclomethasone, Placebo, Ciclesonide
  Arms: 4 Treatment Sequence-Q and B, P and P, A and O
Drug: Placebo/Placebo, Alvesco/Omnaris, QVAR/Beconase — Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID, Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD, QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID
  Other Names: Placebo, Ciclesonide, Beclomethasone
  Arms: 5 Treatment Sequence-P and P, A and O, Q and B
Drug: Placebo/Placebo, QVAR/Beconase, Alvesco/Omnaris — Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID, QVAR Inhalation Aerosol 40 mcg BID and Beconase AQ Nasal Spray 168 mcg BID, Alvesco Inhalation Aerosol 80 BID and Omnaris Nasal Spray 200 mcg QD
  Other Names: Placebo, Beclomethasone, Ciclesonide
  Arms: 6 Treatment Sequence-P and P, Q and B, A and O

SUMMARY:
This study will provide the clinicians guidance on the safest combination of inhaled and nasal corticosteroids for children with mild asthma and allergic rhinitis respectively; however, one safety concern is that these products are independently known to have dose-related effects on short term and intermediate term growth. Knemometry is a non invasive technique for measuring short-term lower leg growth in children and is currently the method of choice in growth studies of short duration. Subjects will be seen on a weekly basis for 18 weeks and at each visit, lower leg length will be measured using knemometry.

DETAILED DESCRIPTION:
This will be a single-center, cross-over study evaluating the effect of Omnaris Nasal Spray 200 mcg QD and Alvesco Inhalation Aerosol 80 BID versus Beconase AQ Nasal Spray 168 mcg BID and QVAR Inhalation Aerosol 40 mcg BID versus Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID on short term growth in pediatric subjects with mild asthma and allergic rhinitis. During the course of the study, subjects will be seen on a weekly basis and lower leg length will be measured using knemometry. Knemometry is a non invasive technique for measuring short-term lower leg growth in children and is currently the method of choice in growth studies of short duration. During the run-in and wash-out periods, subjects will not be treated with any medications or placebos. During the active treatment periods, subjects will be treated with Omnaris Nasal Spray 200 mcg QD and Alvesco Inhalation Aerosol 80 BID or Beconase AQ Nasal Spray 168 mcg BID and QVAR Inhalation Aerosol 40 mcg BID, or Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID. Eligible subjects will be randomized into the study which will contain one run-in period (Period 1), 3 active treatment periods (Periods 2, 4 and 6) and 2 washout periods (Periods 3 and 5). Each period will be of 3 weeks duration and the entire study duration will be 18 weeks. Subjects will be seen on a weekly basis for 18 weeks and at each visit, lower leg length will be measured using knemometry.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will include females and males 6 to 15 years of age.
2. All subjects must have a history of physician diagnosed mild asthma and allergic rhinitis as documented by PCP medical record or detailed history by study investigator.
3. All subjects must have a height within normal limits (5th to 95th percentile) and no history of abnormal growth as assessed by medical history.
4. Subjects may be on current treatment with montelukast as this drug does not affect growth. If a subject is on montelukast at screening/baseline, they will remain on a stable dose throughout the study.
5. Subjects must be willing to comply with study requirements.

Exclusion Criteria:

1. Subjects will be excluded if they have asthma greater than mild persistent severity as defined by NHLBI guidelines.

2 Subjects will be excluded if they used any systemic steroids within the past 60 days.

3. Subjects will be excluded if they had more than one burst of systemic steroids within the past year.

4. Subjects will be excluded if their baseline FEV1 is < 80% predicted. 5. Subjects will be excluded if they have any other serious systemic disease other than asthma.

6. Subjects will be excluded if they have taken any medication known to affect growth i.e. ADHD medications within the past 60 days 7. Subjects will be excluded if they have a history of allergy to any of the study medications.

8. Subjects will be excluded if they have active chickenpox or measles or recent exposure to chickenpox or measles.

9. Subjects will be excluded if they have any history of tuberculosis of the respiratory tract.

10. Subjects will be excluded if they have any active fungal, bacterial, viral or parasitic infections.

11. Subjects will be excluded if they have any history of herpes simplex infection of the eye.

12. Subjects will be excluded if they have taken any immunosuppressive drugs within the past 2 months.

13. Subjects will be excluded if they have any history of Churg-Strauss syndrome or other eosinophilic disorders.

14. Subjects will be excluded if an investigator deems they have any mental or development health issues, such as autism, moderate to severe mental retardation or severe ADHD, that interferes with their ability to complete the knemometry measurements.

15. Subjects will be excluded if an investigator deems they have any physical issues, such as inability to sit independently or amputation of lower leg, that interferes with their ability to complete the knemometry measurements.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Gentile, MD, Principal Investigator — Allegheny General Hospital/Allegheny Singer Research Institute
Locations (2):
- United States (2):
  - Pediatric Alliance-Greentree Division, Green Tree, Pennsylvania
  - Alleghney General Hospital, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- A and O, Then Q and B, Then P and P: Treatment Order: Alvesco and Omnaris; QVAR and Beconase; Placebo and Placebo
- A and O, Then P and P, Then Q and B: Treatment Order: Alvesco and Omnaris; Placebo and Placebo; QVAR and Beconase
- Q and B, Then A and O, Then P and P: Treatment Order: QVAR and Beconase; Alvesco and Omnaris; Placebo and Placebo
- Q and B, Then P and P, Then A and O: Treatment Order: Qvar and Beconase; Placebo and Placebo; Alvesco and Omnaris
- P and P, Then A and O, Then Q and B: Treatment Order: Placebo and Placebo; Alvesco and Omnaris; Qvar and Beconase
- P and P, Then Q and B, Then A and O: Treatment Order: Placebo and Placebo; Qvar and Beconase; Alvesco and Omnaris
Period: Run-In Period (3 Weeks)
Arm/Group | A and O, Then Q and B, Then P and P | A and O, Then P and P, Then Q and B | Q and B, Then A and O, Then P and P | Q and B, Then P and P, Then A and O | P and P, Then A and O, Then Q and B | P and P, Then Q and B, Then A and O
Started | 3 | 4 | 3 | 4 | 4 | 4
Completed | 3 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Treatment Period (3 Weeks)
Arm/Group | A and O, Then Q and B, Then P and P | A and O, Then P and P, Then Q and B | Q and B, Then A and O, Then P and P | Q and B, Then P and P, Then A and O | P and P, Then A and O, Then Q and B | P and P, Then Q and B, Then A and O
Started | 3 | 4 | 3 | 4 | 4 | 4
Completed | 3 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Wash Out Period (3 Weeks)
Arm/Group | A and O, Then Q and B, Then P and P | A and O, Then P and P, Then Q and B | Q and B, Then A and O, Then P and P | Q and B, Then P and P, Then A and O | P and P, Then A and O, Then Q and B | P and P, Then Q and B, Then A and O
Started | 3 | 4 | 3 | 4 | 4 | 4
Completed | 3 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Treatment Period (3 Weeks)
Arm/Group | A and O, Then Q and B, Then P and P | A and O, Then P and P, Then Q and B | Q and B, Then A and O, Then P and P | Q and B, Then P and P, Then A and O | P and P, Then A and O, Then Q and B | P and P, Then Q and B, Then A and O
Started | 3 | 4 | 3 | 4 | 4 | 4
Completed | 3 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Wash Out Period (3 Weeks)
Arm/Group | A and O, Then Q and B, Then P and P | A and O, Then P and P, Then Q and B | Q and B, Then A and O, Then P and P | Q and B, Then P and P, Then A and O | P and P, Then A and O, Then Q and B | P and P, Then Q and B, Then A and O
Started | 3 | 4 | 3 | 4 | 4 | 4
Completed | 3 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Period: Third Treatment Period (3 Weeks)
Arm/Group | A and O, Then Q and B, Then P and P | A and O, Then P and P, Then Q and B | Q and B, Then A and O, Then P and P | Q and B, Then P and P, Then A and O | P and P, Then A and O, Then Q and B | P and P, Then Q and B, Then A and O
Started | 3 | 4 | 3 | 4 | 4 | 3
Completed | 3 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Wash Out Period (3 Weeks)
Arm/Group | A and O, Then Q and B, Then P and P | A and O, Then P and P, Then Q and B | Q and B, Then A and O, Then P and P | Q and B, Then P and P, Then A and O | P and P, Then A and O, Then Q and B | P and P, Then Q and B, Then A and O
Started | 3 | 4 | 3 | 4 | 4 | 3
Completed | 3 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Omnaris Nasal Spray & Alvesco Inhalation Aerosol vs Beconase AQ Nasal Spray & QVAR Inhalation Aerosol on Short-term Lower Leg Growth Velocity as Measured by Knemometry in Pediatric Subjects w/ Mild Asthma & Allergic Rhinitis.
Description: To evaulate the effect of Omnaris Nasal Spray 200 mcg QD and Alvesco Inhalation Aerosol 80 BID versus Beconase AQ Nasal Spray 168 mcg BID and QVAR Inhalation Aerosol 40 mcg BID on- short-term lower leg growth as measured by knemometry in children with mild asthma and allergic rhinitis.
Time Frame: 1 yr
Measure: Mean (95% Confidence Interval); unit: mm/wk
Arm/Group | Alvesco and Omnaris | Beconase and QVAR
Number analyzed (Participants) | 21 | 22
mm/wk | 0.23 [0.04 to 0.41] | 0.33 [0.14 to 0.51]

2. Secondary Outcome: The Effects of Omnaris Nasal Spray & Alvesco Inhalation Aerosol vs Placebo Nasal Spray & Placebo Inhalation Aerosol on Short-term Lower Leg Growth Velocity as Measured by Knemometry in Pediatric Subjects w/ Mild Asthma & Allergic Rhinitis.
Description: To evaluate growth suppressive effect of Omnaris Nasal Spray 200 mcg QD and Alvesco Inhalation Aerosol 80 BID as compared to Placebo Nasal Spray QD and Placebo Inhalation Aerosol BID on short-term lower leg growth velocity as measured by knemometry in children with mild asthma and allergic rhinitis.
Time Frame: 1 yr
Measure: Mean (95% Confidence Interval); unit: mm/wk
Arm/Group | Omnaris & Alvesco | Placebo & Placebo
Number analyzed (Participants) | 21 | 22
mm/wk | 0.23 [0.04 to 0.41] | 0.51 [0.32 to 0.70]

ADVERSE EVENTS:
Arm/Group | Alvesco and Omnaris | Qvar and Beconase | Placebo and Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 7/21 | 7/22 | 6/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alvesco and Omnaris (N=21) | Qvar and Beconase (N=22) | Placebo and Placebo (N=22)
Headaches/migraine (General disorders) | 5 | 4 | 5
Respiratory infections (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 4
Sinus infection (General disorders) | 1 | 1 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Foot pain during sports (General disorders) | 0 | 1 | 1
Swollen eyelid and adenopathy (Eye disorders) | 1 | 0 | 0
Sprained ankle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Viral gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0
Impetigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Bilateral otitis media (Ear and labyrinth disorders) | 1 | 0 | 0
Mouth pain (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No